CLINICAL TRIAL: NCT00203164
Title: A Bi-national, Multicenter, Double-Blind, Randomized Study to Evaluate the Safety and Tolerability of Rasagiline Mesylate in Advanced Parkinson's Disease (PD) Patients With Motor Fluctuations Treated With Chronic Levodopa/Carbidopa Therapy
Brief Title: Study to Evaluate the Safety and Tolerability of Rasagiline in Advanced Parkinson's Disease Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Siyu Liu, MD, PhD, VP IRD, Head of Global Clinical Operations, Teva Branded Pharmaceutical Products IR&D
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVP - 1012/135 Open Label
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rasagiline mesylate (Experimental): rasagiline mesylate 1 mg oral once daily
  Interventions: Drug: rasagiline mesylate

INTERVENTIONS:
Drug: rasagiline mesylate — rasagiline mesylate 1 mg oral once daily

SUMMARY:
This is a study to look at the effectiveness, tolerability, and safety of one dose of rasagiline in advanced Parkinson's disease (PD) patients who have been treated with Levodopa/Carbidopa therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed the Week 26 visit of TVP 1012/133 (Visit 06) in accordance with the protocol.
* Women must be postmenopausal, surgically sterile, or using adequate birth control methods. Women of childbearing potential must have a negative pregnancy test at Baseline/Month 0.
* Patients must be willing and able to give informed consent.

Exclusion Criteria:

* Serious or severe, test drug-related (probable or definite) adverse reaction in study TVP 1012/133.
* Premature discontinuation from study TVP 1012/133 for any reason.
* A clinically significant or unstable medical or surgical condition which would preclude safe and complete study participation. Such conditions may include cardiovascular, pulmonary, hepatic, renal, or metabolic diseases; or malignancies, as determined by medical history, physical exam, skin evaluation, laboratory tests, chest x-ray, or electrocardiogram (ECG).

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2002-05; Primary Completion 2005-07 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
long-term safety and tolerability of rasagiline or levodopa/benserazide (LD/BZD) therapy | until commericially available
  To evaluate the long-term safety and tolerability of rasagiline in PD patients with motor fluctuations treated with chronic levodopa/carbidopa (LD/CD) or levodopa/benserazide (LD/BZD) therapy

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Salzman, Ph.D., Study Director — Teva Neuroscience, Inc.
Locations (6):
- United States (6):
  - Margolin Brain Institute, Fresno, California
  - Rush - Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Creighton University, Omaha, Nebraska
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania